CLINICAL TRIAL: NCT05623735
Title: Comparison of the Effects of Two Different Instrument Assisted Soft Tissue Mobilization Techniques in Individuals With Chronic Non-Specific Low Back Pain
Brief Title: Comparison of the Effects of Instrument Assisted Soft Tissue Mobilization Techniques Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ETK00-2022-0173
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Chronic Low-back Pain
Keywords: IASTM; chronic pain; flexibility; disability; mobility; muscular endurance
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrument Assisted Soft Tissue Mobilization (IASTM) Group While Lying Prone (Experimental): The application will take a total of 6 sessions, with two sessions per week for 3 weeks.
  While individuals are lying in the prone position, the IASTM protocol will be applied bilaterally on the erector spinae and then on the hamstrings. The application will take approximately 17 minutes.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization Group While Lying Prone
- Instrument Assisted Soft Tissue Mobilization Group Combined with Functional Movement (Experimental): While standing in the "extended child pose (utthita balasana)" stance, the "IASTM" protocol will be applied bilaterally on the lumbar erector spines, with the hands on them and moving back to the old position. Then, the "IASTM" protocol will be applied bilaterally on the hamstrings by making consecutive knee flexion-extension up to 90 degrees while the individuals are lying prone.
  The application will take approximately 17 minutes.
  Interventions: Other: Instrument Assisted Soft Tissue Mobilization Group Combined with Functional Movement

INTERVENTIONS:
Other: Instrument Assisted Soft Tissue Mobilization Group While Lying Prone — 1. Sliding movements in all directions at 30 - 60 degree angles will be made in the form of mobilizations of 45 seconds with instruments.
  2. Mobilizations of 45 seconds will be made with instruments along the quarter circle line in all directions at 30 - 60 degree angles.
  3. Starting with an angle of 60 degrees on the area to be treated, the movement of shifting towards an angle of 30 degrees will be made in all directions for 30 seconds.
  4. The tissue will be mobilized for 30 consecutive seconds, starting from just caudal to your waist and drawing the letter J towards the cranial.
  5. Sliding movements in all directions at 30 - 60 degree angles will be made with instruments in the form of mobilizations for 45 seconds.
  6. Mobilizations of 45 seconds will be made with instruments along the quarter circle line in all directions at 30 - 60 degree angles.
  7. 30 - 60 degree swipe movement shorter brushing style small movements will be done for 30 seconds.
  Arms: Instrument Assisted Soft Tissue Mobilization (IASTM) Group While Lying Prone
Other: Instrument Assisted Soft Tissue Mobilization Group Combined with Functional Movement — 1. Sliding movements in all directions at 30 - 60 degree angles will be made in the form of mobilizations of 45 seconds with instruments.
  2. Mobilizations of 45 seconds will be made with instruments along the quarter circle line in all directions at 30 - 60 degree angles.
  3. Starting with an angle of 60 degrees on the area to be treated, the movement of shifting towards an angle of 30 degrees will be made in all directions for 30 seconds.
  4. The tissue will be mobilized for 30 consecutive seconds, starting from just caudal to your waist and drawing the letter J towards the cranial.
  5. Sliding movements in all directions at 30 - 60 degree angles will be made with instruments in the form of mobilizations for 45 seconds.
  6. Mobilizations of 45 seconds will be made with instruments along the quarter circle line in all directions at 30 - 60 degree angles.
  7. 30 - 60 degree swipe movement shorter brushing style small movements will be done for 30 seconds.
  Arms: Instrument Assisted Soft Tissue Mobilization Group Combined with Functional Movement

SUMMARY:
The aim of this study is to determine whether the effectiveness of instrument-assisted soft tissue mobilization technique is different from passive prone lying when performed with a functional exercise in individuals with chronic nonspecific low back pain.

DETAILED DESCRIPTION:
Individuals participating in the study will first be divided into two groups by randomization. While IASTM (Instrument Assisted Soft Tissue Mobilization Techniques) will be applied to one group in the prone position, IASTM will be applied to the other group with functional exercise. The pain, mobility, flexibility, disability and endurance parameters of the individuals assigned to the groups after randomization will be determined just before the application, immediately after the 1st application and immediately after the 6th application. The study will last for a total of 6 sessions, with two sessions per week for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with non-specific low back pain by a specialist physician
* 18-45 years old
* Having 3 or more pains on VAS for the last 3 months.
* Those who do not use analgesic drugs
* Not taking physiotherapy for the last 6 months.

Exclusion Criteria:

* Those with orthopedic, neurological, psychiatric and systemic diseases (such as fracture, osteoporosis, scoliosis, kyphosis, stenosis, cauda equina, myositis ossificans, severe nerve compressions, rheumatoid arthritis, cancer)
* Those with a history of spinal surgery
* Pregnant and lactating
* Open wound, infection, serious kidney disease
* Those who have limited hip joint movements

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 3 Weeks
  Individuals' pain levels will be measured using the Visual Analogue Scale (VAS) both at rest and during activity. It will be requested to mark any point on a horizontal line of 10 cm length such that 0 no pain, 10 unbearably severe pain.

SECONDARY OUTCOMES:
Mobility (Modified Schober Test) | 3 Weeks
  Individuals' spinal mobility will be assessed using the Modified Schober Test. While the patient is standing, the midpoint between the spina iliaca posterior superior is marked. This point is considered the L4-L5 level. Two more points are marked 10 cm above and 5 cm below this point. This distance will be measured both while standing and by asking them to bend forward without bending the knees, with the hands touching the feet.
Flexibility (Sit and Reach Test) | 3 Weeks
  A measuring bench with a length of 55 cm in the upper part, 35 cm in the lower part, 32 cm in height and 45 cm in width will be used. The soles of both lower extremities will be fully touching the bench with bare feet and the patient will be asked to lie on the bench with knees extended straight and hands on top of each other. The level of the feet will be the 0 point on the table at the top. It will be recorded in such a way that it extends forward +, lagging behind -. The test will be calculated by taking the best value of the measurements after 3 consecutive repetitions.
Flexibility (Maximal Hip Flexion Active Knee Extension (MHFAKE)) | 3 Weeks
  Hamstring flexibility will be measured using the Active Knee Extension Test with Maximal Hip Flexion (MHFAKE). It has been reported to be the best measure of hamstring flexibility compared to traditional straight leg raises or other tests. While the individual is lying in the supine position, he will be asked to take the hip of the tested extremity to its maximal flexion and lock it with his hands, then actively bring the knee to the extension position until it reaches the maximal tension it can reach. The contralateral limb will be extended straight on the bed. To prevent variations, the contralateral extremity will be fixed to the bed from the distal thigh with a belt. Knee angle will be measured with a goniometer.
Disability (Oswestry Disability İndex) | 3 Weeks
  The Turkish version of the Oswestry Low Back Pain Disability Questionnaire consisting of 10 questions will be used in order to measure the loss of function caused by low back pain. These questions are; It consists of questions compatible with daily life activities such as pain intensity, personal care, lifting/carrying, walking, sitting, standing, sleep, travel, social life, and degree of pain change. Higher scores mean more disability.
Trunk Extensors Muscle Endurance (Biering-Sorenson Test) | 3 Weeks
  The trunk extensors muscle endurance of individuals will be evaluated with the Biering Sorenson test. Individuals will be asked to lie face down on the bed and extend their torso out of the bed from the anterior superior iliac spine (SIAS). A rolled towel will be placed in front of the ankle and their legs will be supported by the physiotherapist. Individuals will be asked to stand with their hands crossed in the pectoral region and keep their torso parallel to the ground against gravity. The time will be recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Süleyman Güzelşemme, Res. Asst., Principal Investigator — Eastern Mediterranean University; Sevim Öksüz, Asst. Prof., Study Director — Eastern Mediterranean University
Locations (1):
- Süleyman Güzelşemme, Famagusta, Cyprus